CLINICAL TRIAL: NCT06184022
Title: Augmented Reality Serious Game Design for Promoting Children's Science Education Cognition: a Randomized Controlled Trial
Brief Title: Augmented Reality Serious Game Design for Promoting Children's Science Education Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, zhudian, Dr, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sjtu0009
Record Dates: First submitted 2023-12-06; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Educational Problems; Augmented Reality; Serious Game
Keywords: augmented reality; serious game; science education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented reality serious game (Experimental): Before the test started, the experimenter gave the basic information of the experiment to the participants. The participants were requested to complete a cognitive exam on the notion of light, and were asked to perform a POE test for each question. The experimental group utilized the three game lesson modules of the AR science education app designed for this study, including "Animals vision," " Light transmission," and "Color-Light mixing". On their initial encounter with the game, respondents were given around 10 minutes to comprehend its mechanics. The experimental group's total learning time was limited to 20 minutes, the testing process was completed under the supervision of the instructor and the experimenter. During the experiment, the participants were not disturbed in any way; researchers only intervened when they faced difficulties or requested assistance. The participants were given a 15-minute respite at the conclusion of the trial to take another POE test.
  Interventions: Combination Product: Augmented reality serious game design for promoting children's science education cognition:
- non-ar serious game (Active Comparator): The control group completed the same three game courses for a maximum of 20 minutes using the non-AR app "Light and Color" after completing the pre-test.For the non-AR game we used "Light and Color" designed by Tinybop available in Appstore Tools for young artists and scientists. Both games have the same scientific educational content on optics (in fact, to experiment with control variables, we adopted the same scientific knowledge as in this non-AR app at the stage of designing the content), so it is possible to perform a POE test. The participants took a 15-minute break at the conclusion of the trial to complete another POE test and the IMI scale.
  Interventions: Combination Product: Augmented reality serious game design for promoting children's science education cognition:

INTERVENTIONS:
Combination Product: Augmented reality serious game design for promoting children's science education cognition: — The experimental group utilized the three game lesson modules of the AR science education app designed for this study, including "Animals vision," " Light transmission," and "Color-Light mixing".
  The experimental group's total learning time was limited to 20 minutes, the testing process was completed under the supervision of the instructor and the experimenter, and the children's behavioral characteristics were recorded. During the experiment, the participants were not disturbed in any way; researchers only intervened when they faced difficulties or requested assistance. The participants were given a 15-minute respite at the conclusion of the trial to take another POE test. Before and after the intervention, each participant's performance on the game was recorded.
  Other Names: AR serious game

SUMMARY:
Background：The process of constructing knowledge in the context of children's science education plays a significant role in fostering the development of early scientific literacy. Nevertheless, children sometimes struggle to comprehend scientific knowledge due to the presence of abstract notions.

Objective: To evaluate the efficacy of augmented reality (AR) games as a teaching tool for enhancing children's understanding of optical science education.

Methods: 36 healthy children between the ages of 6 and 8 years old were included in this study. Individuals were randomly divided into an intervention group (n=18) and a control group (n=18). Interventions, namely a 20-minute AR science education including three game lesson modules, while the control group was asked to learn 20-minute same knowledge with non-AR science learning app. POE (predict-observe-explain) test of 3 games including animal vision, color-light mixing and light refraction were conducted for all participants before and after the experiment. Also, intrinsic Motivation Inventory (IMI) test including interest-enjoyment (INT-ENJ), perceived competence (COMP), effort-importance (EFF-IMP), and tension-pressure (TEN-PRESS) were conducted for children after the experiment.

DETAILED DESCRIPTION:
Guardians of children with independent mobility provided informed written consent for their participation in the study. Participants were randomly assigned to the experimental and control groups using a randomization list maintained by members of the study group uninvolved in any other aspect of the research. Participants' guardians received and opened opaque, sealed envelopes containing group assignments following the initial evaluation. The evaluator in charge of assessing the results of the AR scientific education course had no access to participant information or group assignment.

Sample size calculations were performed using PASS based on the POE test scores from the pre-experiment. Group sample sizes of 18 and 18 achieve 90.118% power to reject the null hypothesis of equal means when the population mean difference is μ1 - μ2 = 3.2- 1.0 = 2.2 with a standard deviation (SD) for two groups of 2.0 and 1.9, and with a significance level (a) of 0.050 using a bilateral, two-sample, equal-variance t-test.

This experiment was a randomized controlled trial, and the participants were randomly separated into the experimental group and the control group. The random numbers were generated by applying SAS software analysis system on computer simulation, and no experimental group was allowed to be selected at random. Every child was tested in the company of a guardian and two experimentalists.

The independent variable was the type of game ("Light and Color", a light science educational product and AR game we designed). The independent variable was the type of game ("Light and Color", a light science educational product and AR game that we created). The dependent variables for both experimental and control group students were the difference between the pre- and post-test results of the POE test and the children's motivation to play the game. To create control variables for the experiment, both games were based on animal vision, light transmission, and color-light mixing, and neither game involved the teacher. In addition, there were no significant gender or age differences between the two student groups.

ELIGIBILITY:
Inclusion Criteria:

* native Chinese children (6-8 years old)
* Clear cognition

Exclusion Criteria:

* Poor listening and comprehension abilities

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
POE (predict-observe-explain) test | 30 minutes
  The POE (predict-observe-explain) test is commonly used in science classes and tries to expose students' expectations about certain events and the rationale for these predictions [19]. It is used to demonstrate scientific experiments to pupils and is advantageous for fostering children's critical thinking and assessing students' grasp of scientific topics. The investigator then displays the relevant physical events to the students using basic prop materials after requiring the students to independently determine the questionnaire's responses and their justifications. Finally, students were instructed to alter or supplement their explanations in light of the observations.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) | 30 minutes
  It was developed under game conditions with three subscales [22]: interest-enjoyment (INT-ENJ), perceived competence (COMP), and effort-importance (EFF-IMP) to assess the perceived levels of motivation, enjoyment, and perceived difficulty of the participants. To investigate the negative emotions of children using the AR, the study inserted questions from the original scale's tension-stress section

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Liu, Prof, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Dian Zhu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
If necessary, the data can be obtained by contacting the author.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: After the paper is accepted.
Access Criteria: zhudian@sjtu.edu.cn